CLINICAL TRIAL: NCT01658241
Title: A Phase II Study to Investigate Biological Correlates of Clinical Response to Panobinostat in Haematological Malignancy
Brief Title: Panobinostat Biological Correlates Study
Acronym: VEG VCA1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12/18
Record Dates: First submitted 2012-07-20; First posted 2012-08-06 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Nodal Lymphoma; Lymphoma With Cutaneous Involvement; Lymphoma in Leukemic Phase; Marrow Involvement With Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Main population (Experimental)
  Interventions: Drug: panobinostat

INTERVENTIONS:
Drug: panobinostat — 40mg, three times a week, oral pill over 12 cycles, 4 weeks per cycle
  Other Names: LBH589

SUMMARY:
This study is looking at the effects of Panobinostat, an investigational treatment, on cancer cells in patients who have Hodgkin lymphoma (a cancer of the immune system with specific Hodgkin/Reed Sternberg Cells), T-cell lymphoma (a cancer of the immune system with too many T lymphocytes), chronic lymphocytic leukemia or prolymphocytic leukaemia (immune system with too many lymphocytes in the blood stream), lymphoplasmacytic lymphoma (immune system with too many plasma cells or B lymphocytes) or myeloma (a cancer of plasma cells).

Panobinostat is a new drug which has led to disease improvement in some patients with Hodgkin lymphoma, certain types of T-cell lymphoma, myeloma and some B cell lymphomas. Not all patients benefit from panobinostat.

The researchers wish to look at the effects of panobinostat on cancer cells. The aim of this project is find out which patients or diseases are likely to respond to treatment with panobinostat in the future and to see if there are particular features of the patient or of the cancer that affects the likelihood of the way individuals respond to panobinostat.

Panobinostat is an oral medication (taken by mouth) that effects the way cancer cells and in normal cells make proteins. Panobinostat has been used in several clinical trials around the world. The largest trials generally have fewer than 200 patients and are in Hodgkin lymphoma, cutaneous T-cell lymphoma, and myeloma where between one in five and one in three patients have significant improvement in their disease.

Researchers will look at samples of tumour before treatment and during treatment. This will be one of the first studies to look at how cancer cells change following treatment with this drug. It is unusual because it requires repeated biopsies of the participant's tumour. Panobinostat is considered an experimental (or investigational) drug and not approved by any regulatory authority (such as the Food and Drug Administration, FDA in the USA or by the Therapeutics Goods and Administration, TGA, in Australia) to treat any type of cancer. Therefore, Panobinostat is not approved to treat patients who have been diagnosed with refractory or relapsed cancer.

A total of 30 patients with one of the diseases listed above will be enrolled at Peter MacCallum Cancer Centre.

It is expected it will take about 2 to 3 years to recruit 30 patients and that on average patients will take part for six to eighteen months. This time could be shorter or longer depending on how well the treatment works in each individual. While the trial will take up to 4 years to complete, the science studies may take longer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven lymphoproliferative neoplasm belonging to one of the following disease categories that has relapsed or has an incomplete response to conventional therapy, or where the patient is considered intolerant to conventional chemotherapy or where no other conventional therapy is considered appropriate.

   * Hodgkin lymphoma
   * Multiple myeloma (patient must have been exposed to or otherwise unable to tolerate lenalidomide and bortezomib).
   * Peripheral T-cell lymphoma (including angioimmunoblastic lym-phoma and PTCL Not otherwise specified)
   * Cutaneous T-Cell lymphoma [Mycosis fungoides, Sézary syndrome, Primary cutaneous gamma-delta T cell lymphoma, Lymphomatoid papulosis, Subcutaneous panniculitis-like T cell lymphoma Alpha/Beta or lambda/delta type and CD30+ Anaplastic large cell lymphoma]
   * Cutaneous B-cell lymphoma [Extranodal marginal zone lymphoma of mucosa-associated lymphoid tissue (MALT) lymphoma of the skin, Primary cutaneous follicle cell lymphoma, Primary cutaneous DLBCL, leg type]
   * Chronic lymphocytic leukaemia
   * Lymphoplasmacytic lymphoma
   * B-prolymphocytic leukaemia (or CLL in prolymphocytic transfor-mation)
   * T-prolymphocytic leukaemia
2. The lymphoma needs to be accessible, convenient and safe (< 5% risk of bleeding or serious event) for biopsy in at least one of the following sample types on multiple occasions as stipulated by the study protocol:

   * Peripheral blood samples (absolute peripheral circulating lymphoma cells > 2x109/L).
   * Bone marrow biopsy (> 30% marrow involvement by lymphoma).
   * Clinically apparent cutaneous lymphoma amenable to skin biopsy (patients with cutaneous involvement and blood stream involvement must agree to biopsies of the skin in addition to peripheral blood samples).
   * Clinically accessible lymph node or extranodal disease amenable to core biopsy.
3. Age ≥ 18 years
4. ECOG performance status score 0-2 at screening.
5. Life expectancy of ≥12 weeks
6. Patient has the following laboratory values within 3 weeks of starting study drug (labs may be repeated, if needed, to obtain acceptable values before failure at screening is concluded)

   * ANC ≥ 1.5x109 /L
   * Platelet count ≥ 100 x 109 /L (unless due to marrow involvement)
   * AST/SGOT and ALT/SGPT ≤ 2.5 x ULN
   * Serum total bilirubin ≤ 1.5 x ULN (except gilbert's syndrome, in which case ≤ 3 x ULN is required)
   * Serum creatinine ≤ 1.5 x ULN
   * Serum potassium, magnesium, phosphorus, sodium, total calcium (corrected for serum albumin) or ionized calcium within normal limits
7. Patient has the ability to swallow capsules.
8. Sexually active patient (men and women of child bearing potential) agrees to use double barrier method of contraception during the course of the study treatment period (13 cycles) and for 3 months after completing study treatment. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who are not postmenapausal (no menses) for at least 12 consecutive months.
9. Males with a female partner of childbearing potential must agree to use a medically reliable method of preventing conception throughout the study and for 30 days following the date of last dose.
10. Mentally competent and is able to understand the information given and provide informed consent to both the clinical aspects of the study as well as the demands of the correlative studies and associated tumour biopsies.

Exclusion Criteria:

1. Concomitant use (within 28 days of first biopsy) of any anti-cancer therapy including radiation therapy
2. Exposure to a histone deacetylase inhibitor within the preceding 4 weeks.
3. Patient has received chemotherapy or any investigational drug or undergone major surgery ≤ 2 weeks prior to starting study drug or whose side effects of such therapy have not resolved to ≤ grade 1 (except for grade 2 neuropathy).
4. Current involvement (medication delivered within 28 days of first biopsy)in a study of an alternative investigational agent.
5. Impaired cardiac function including any one of the following:

   * LVEF < the lower limit of institutional normal, as determined by ECHO or MUGA
   * Obligate use of a permanent cardiac pacemaker
   * Congenital long QT syndrome
   * History or presence of ventricular tachy-arrhythmias
   * Resting bradycardia defined as < 50 beats per minute
   * QTcF > 450 msec on screening ECG
   * Complete left bundle branch block, bifasicular block
   * Any clinically significant ST segment and/or T-wave abnormalities
   * Presence of unstable atrial fibrillation (ventricular rate > 100 bpm). Patient with stable atrial fibrillation is allowed in the study provided the other cardiac exclusion criteria are satisfied.
   * Myocardial infarction or unstable angina pectoris ≤ 6 months prior to starting study drug
   * Congestive heart failure (New York Heart Association class III-IV)
   * Other clinically significant heart disease and vascular disease (e.g. uncontrolled hypertension)
6. Patient is taking medications with relative risk of prolonging the QT interval or inducing torsade de pointes, if such treatment cannot be discontinued or switched to a different medication prior to starting study drug
7. Patient has impairment of GI function or GI disease that may significantly alter the absorption of panobinostat, such as:

   * Active ulcerative disease
   * uncontrolled nausea or vomiting
   * diarrhea CTCAE grade ≥ 2 (despite antidiarrheal medications)
   * malabsorption syndrome
   * obstruction
   * stomach and/or small bowel resection
8. Known HIV, hepatitis B or hepatitis C (a screening test is not required)
9. Female patients who are pregnant or breast feeding
10. Other concurrent severe and/or uncontrolled medical conditions such as (but not limited to)

    * uncontrolled diabetes
    * active or uncontrolled infection
    * chronic obstructive or chronic restrictive pulmonary disease including dyspnea at rest from any cause
    * uncontrolled thyroid dysfunction
    * recent, acute or active bleeding
11. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule. This condition must be discussed with the patient prior to signing consent and registration in the trial.
12. Prior diagnosis of cancer that was:

    * more than 3 years prior to current diagnosis with subsequent evidence of disease recurrence or estimated clinical expectation of recurrence is greater than 10% within next 2 years
    * within 3 years of current diagnosis with the exception of successfully treated basal cell or squamous cell skin carcinoma, carcinoma in situ of the cervix or localised cancer treated curatively with local therapy only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07-16 (Actual); Primary Completion 2015-03-18 (Actual); Study Completion 2015-03-18 (Actual)

PRIMARY OUTCOMES:
Change in gene expression profile of tumor samples taken before and after treatement with panobinostat | Up to two years from trial entry

SECONDARY OUTCOMES:
Overall response (OR): this is a composite clinical endpoint including those who have achieved a complete remission (CR) or partial remission (PR) by conventional disease-appropriate criteria. (i.e. OR=CR+PR) | Up to two years from trial entry
Clinical benefit: a composite endpoint including those with complete remission, partial remission, marginal response and those with otherwise stable disease that has been maintained for at least 2 cycles of therapy | Up to two years from trial entry
Time to response: the time from first drug dose to best confirmed response | Up to two years from trial entry
Time to progression: the time from initial observation of response to confirmed disease progression, or the time from first drug dose to confirmed disease progression | Up to two years from trial entry
Progression-free survival: time from trial registration to disease progression or death from any cause | Up to two years from trial entry
Disease-specific biological improvement - as defined in the protocol | Up to two years from trial entry
Sustained disease-specific biological improvement - as defined in the protocol | Up to two years from trial entry

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dickinson, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia